CLINICAL TRIAL: NCT05173753
Title: Novel Self-Adhesive Composite Hybrid Versus Conventional Composite in Restoration of Carious Primary Teeth. A Split Mouth Randomized Clinical Trial
Brief Title: Novel Self-Adhesive Composite Hybrid Versus Conventional Composite in Restoration of Carious Primary Teeth.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Fatima Elfadil Rabie, Principal investigator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Surefil one in primary teeth
Record Dates: First submitted 2021-12-04; First posted 2021-12-30 (Actual); Last update posted 2022-07-27 (Actual); Status verified 2022-07

CONDITIONS: Dental Caries in Children

STUDY DESIGN:
Intervention Model Description: for both the intervention group and control group, the procedure and follow up will be done parallel to each other(same time).
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Novel self-adhesive composite restoration (Surefil one) (Active Comparator)
  Interventions: Other: Novel self-adhesive hybrid composite(Surefil one)
- conventional composite resin restoration(VOCO Grandio) (Active Comparator)
  Interventions: Other: Novel self-adhesive hybrid composite(Surefil one)

INTERVENTIONS:
Other: Novel self-adhesive hybrid composite(Surefil one) — Surefil one, is a recent introduced esthetic dental restoration for treatment of carious teeth.

SUMMARY:
The clinical trial aim to evaluate clinical effectiveness of self-adhesive composite hybrid (Surefil one) versus conventional composite(VOCO Grandio) as restorative material for carious primary teeth.

DETAILED DESCRIPTION:
Composite resin is a continuous improving material as its full fill many requirements seeking in dental restorative materials, but is the new introducing composite resin material is always better than the previous one? This randomized clinical trial is performed to discus and assess that hypothesis. A total of 120 class I restoration(60 Surefil one novel self-adhesive composite hybrid & 60 VOCO Grandio conventional composite resin) will be placed in posterior teeth of 60 volunteers(splint mouth design) following the manufacturer instruction. age between 4-7 years. The restorations will then be evaluate clinically at baseline, 3, and 6 month intervene. Both the procedure and follow up will done in the out-patient clinic, Pediatric Dentistry and Dental Public Health Department, Faculty of Dentistry, Cairo University, Cairo, Egypt.

ELIGIBILITY:
Inclusion criteria:

Children:

Good general health and medically free patients. Age ranges: from 4-7 years old. A provided informed consent by the parents. Acceptable child cooperation.

Teeth:

Class I carious primary teeth. 2 contralateral or adjacent carious teeth. Simple caries, extending to the dentin. No singe or symptom of pulp inflammation. Normal radiographic examination.

Exclusion Criteria:

Children:

Unable to attend follow-up visits. Refusal of participation.

Teeth:

Symptom tooth. Periapical Pathosis. Mobile primary tooth.

Ages: 4 Years to 7 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 60 (Estimated)
Dates: Start 2022-08 (Estimated); Primary Completion 2022-12 (Estimated); Study Completion 2023-06 (Estimated)

PRIMARY OUTCOMES:
clinical effectiveness | 6 month intervene
  The two materials will be evaluated using the FDI World Federation criteria.

SECONDARY OUTCOMES:
The cost effectiveness | 6 month intervene
  will be measured using the ICER (Incremental cost-effectiveness ratio)
Duration of procedure | 6 month intervene
  measure using stop watch
Child cooperation | 6 month intervene
  Wright Modification of Frankl behavior scale will be use(Rating1-5 as R1 definitely negative, and R5 definitely positive).

CONTACTS AND LOCATIONS:
Overall Officials: Kamal Aldin El Motayam, Professor, Study Director — Cairo University; Passant Nagi, PHD, Study Director — Cairo University; Mahitab M Abdel khalek, BDS, Principal Investigator — Cairo University; Fatema H Mohamed, BDS, Principal Investigator — Cairo University

IPD SHARING:
Plan to Share IPD: Undecided